CLINICAL TRIAL: NCT05956327
Title: Insight Into Hippocampal Neuroplasticity in Schizophrenia by Investigating Molecular Pathways During Physical Training
Acronym: BrainTrain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Lena Deller, Doctoral Candidate, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BI 576/9-1, FA 241/21-1
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Neuronal Plasticity; Exercise
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Pliability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Aerobic endurance training on a bicycle ergometer
  Interventions: Procedure: Aerobic Endurance Training
- Control Group (Active Comparator): Flexibility, strengthening and balance training
  Interventions: Procedure: Flexibility, strengthening and balance training

INTERVENTIONS:
Procedure: Aerobic Endurance Training — Aerobic endurance training on a bicycle ergometer (week 1 to 6: three units per week á 40 minutes, week 7 to 12: three units á 45 minutes, in groups of up to three patients over 13 weeks)
  Arms: Intervention Group
Procedure: Flexibility, strengthening and balance training — Flexibility, strengthening and balance training (exercises from the areas of stretching, strength, balance and relaxation, 3x40 min from week 1-2, 3x45 min from week 3-4 and 3x50 min from week 5-13, in groups of up to three patients over 13 weeks)
  Arms: Control Group

SUMMARY:
Aerobic endurance training has shown positive effects on symptoms, cognition, daily functioning, and the structure of the hippocampus in patients with schizophrenia. The study investigates genetic and epigenetic influences on neuroplastic changes following three months of endurance training. A control group performs flexibility, strength, and balance training. The main objective is to examine the association between a genetic risk score for schizophrenia and volume increase in the CA4/DG region of the hippocampus. Additional goals include examining changes in synapses, brain structure, function, and metabolism, as well as clinical symptoms and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for voluntary study participation.
* Patients with schizophrenia: diagnosis of schizophrenic psychosis according to ICD10 and DSM V,
* Positive And Negative Syndrome Scale (PANSS) total score ≤ 75 before the start of the intervention
* Reliable contraception in women of childbearing age
* Patients must have been treated with individualized medication according to valid treatment guidelines. All antipsychotic substances are allowed, also as depot medication. Treatment with one as well as with two antipsychotic substances is possible. The additional administration of low- and medium-potency antipsychotic substances as on-demand medication for the treatment of agitation and sleep disorders is possible, provided that the daily dosage of 150 CPZ units is not exceeded. The active substance and dose of the individualized antipsychotic medication used to achieve the inclusion criterion of psychopathological symptom remission must be constant for at least 2 weeks before inclusion in the study.

Exclusion Criteria:

* Lack of reliability and sanity (examined by an independent psychiatrist)
* Positive urine drug screen for illicit drugs (except benzodiazepines)
* Acute suicide risk
* Other relevant psychiatric axis-I disorders according to the diagnostic testing procedure (Mini International Neuropsychiatric Interview, MINI)
* Other relevant neurological or other disorders
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hippocampal volume | 13 weeks
  Change in hippocampal subregion cornu ammonis (CA) 4 volume (∆CA4/DG) and its correlation with polygenetic risk factor (PRS)

SECONDARY OUTCOMES:
Cognitive functions | 13 weeks
  verbal memory, working memory, motor speed, verbal fluency, attention and speed of information processing assessed by BACS
Executive functions | 13 weeks
  visual attention and task switching (TMT-A, B), episodic memory with the What-Where-When Test and visuo-spatial short- and long-term memory with the Brief Visuospatial Memory Test-Revised (BVMT-R)
Symptoms severity | 13 weeks
  change over study duration assessed by PANSS, BNSS, CDSS
Functioning in daily life | 13 weeks
  Assessed by SOFAS, GAF, FROGS
Cardiovascular risk factors | 13 weeks
  Aerobic fitness levels (W/kg), body weight, waist circumference, body fat, lipid panel, HbA1c, physical activity as assessed with the IPAQ will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Falkai, Prof. Dr., Principal Investigator — Director of the Department of Psychiatry and Psychotherapy, University Hospital, LMU
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes